CLINICAL TRIAL: NCT03473093
Title: The Effect of Adding Pregabalin to the Analgesic Effect of Intravenous Morphine in Patients With Multiple Fracture Ribs
Brief Title: Oral Pregabalin Effect to the Intravenous Morphine in Multiple Fracture Ribs
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Medhat Mahfouz Eshak, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: pain in multiple fracture ribs
Record Dates: First submitted 2018-03-08; First posted 2018-03-22 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Fracture; Rib, Multiple
MeSH Terms: conditions — Fractures, Bone | interventions — Pregabalin; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- morphine (Active Comparator): This group will receive only morphine infusion (20microgram/kg/h)
  Interventions: Drug: Morphine
- pregabalin (Active Comparator): This group will receive only morphine infusion (20microgram/kg/h) and oral pregabalin (150 mg)
  Interventions: Drug: Pregabalin 150mg; Drug: Morphine

INTERVENTIONS:
Drug: Pregabalin 150mg — One group will receive oral pregabalin with morphine infusion
  Arms: pregabalin
Drug: Morphine — One group will receive morphine infusion 20 microgram/kg/h

SUMMARY:
Determine the effect of using oral pregabalin on the analgesic effects of IV infusion of morphine in patients with multiple fracture ribs.

DETAILED DESCRIPTION:
Blunt chest trauma accounts for a significant proportion of debilitating and life-threatening injuries. Rib fractures are notoriously painful and can lead to prolonged hospitalization,contribute to the development of pneumonia and respiratory failure, and delay outpatient recovery significantly.Flail chest, along with chest wall deformity, the most severe of chest wall injuries, is associated with significant acute morbidity and mortality.Flail chest injury has been associated with a high mortality rates historically and up to 16 % more recently. In-patients with physiologic flail visibly apparent paradoxical chest wall motion leads to inefficient respiratory effort and compression of the lung and diminishes the negative intra thoracic pressure essential for the passive movement of air into the bronchial tree. Atelectasis leads to increased lung resistance and decreased compliance, making the work of breathing much more difficult. Loss of the ability to generate negative intra thoracic pressure with breathing also impairs venous return, a passive process dependent on the negative intra thoracic pressure generated with each breath. In patients without a visible flail segment, i.e., an anatomic or radiologic flail,the physiologic derangements can be similarly destructive.There is mounting evidence that a patient's perception of pain in the early post-injury period is associated with chronic pain development . A recent prospective study of rib fracture patients found that pain and disability at 8 weeks post injury could be predicted by the pain intensity within the first few days after injury . Interestingly, the number of fractures and the bilaterality of fractures were not predictive. Thus, pain management in the early post-injury setting is likely paramount to obtaining a more favorable recovery. Opioids, are traditional first-line therapy for acute rib fracture pain. But because of chronic misuse potential and central desensitization concerns, pain researchers and clinicians are increasingly recommending that opioids be used only in combination with other analgesic modalities such acetaminophen, nonsteroidal anti-inflammatory medication(NSAID), the anticonvulsants gabapentin and pregabalin,and the topical lidocaine patch

ELIGIBILITY:
Inclusion Criteria:

* Adult patients above 18 years old
* ASA [1] and ASA [2]
* mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

* Patient coma scale less than 10
* Impaired kidney functions
* Chronic pain syndromes and patients with chronic opioid use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
decrease pain | one week
  measured by visual analogue score ranged from 0 to 10 with higher numbers are worse than lower numbers

SECONDARY OUTCOMES:
I.C.U stay time | one week
  decrease time

REFERENCES:
- [Background] Cannon RM, Smith JW, Franklin GA, Harbrecht BG, Miller FB, Richardson JD. Flail chest injury: are we making any progress? Am Surg. 2012 Apr;78(4):398-402. PMID 22472394
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962